CLINICAL TRIAL: NCT00365144
Title: A Phase II Trial of Bevacizumab Plus Erlotinib for Patients With Metastatic Gemcitabine-Refractory Pancreatic Cancer
Brief Title: Bevacizumab and Erlotinib in Treating Patients With Metastatic Pancreatic Cancer That Did Not Respond to Previous Treatment With Gemcitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 054511; UCSF-054511; UCSF-H12191-28233-01
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Pancreatic Cancer
Keywords: stage IV pancreatic cancer; adenocarcinoma of the pancreas; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab Plus Erlotinib Hydrochloride (Experimental): A treatment cycle is 21 days:
  bevacizumab 15 mg/kg as a 60-90 min infusion once every 21 days, with erlotinib hydrochloride 150 mg by mouth daily
  Interventions: Biological: bevacizumab; Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab
Drug: erlotinib hydrochloride
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of pancreatic cancer by blocking blood flow to the tumor. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving bevacizumab together with erlotinib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with erlotinib works in treating patients with metastatic pancreatic cancer that did not respond to previous treatment with gemcitabine.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the 6-month overall survival rate in patients with gemcitabine hydrochloride-refractory metastatic pancreatic cancer treated with bevacizumab and erlotinib hydrochloride.
* Determine the safety and toxicity of this regimen in these patients.

Secondary

* Evaluate the objective response rate in these patients.
* Evaluate time to tumor progression in these patients.
* Determine the efficacy of this regimen, in terms of the proportion of patients with ≥ 50% decline in carbohydrate antigen 19-9, also called cancer antigen 19-9 (CA19-9) biomarker, in these patients.
* Obtain sequential measurements of circulating tumor cells (micrometastases) and endothelial cells in serum and correlate these variables with clinical outcomes (in patients enrolled in UCSF site only).

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on day 1 and oral erlotinib hydrochloride once daily on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection at baseline and periodically during study for biomarker/laboratory analysis, including the CA19-9 biomarker. Circulating tumor micrometastases and endothelial cells are also measured in patients enrolled in University of California San Francisco (UCSF) site.

After completion of study treatment, patients are followed at 30 days and at 6 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* Documented extrapancreatic metastases

  * Radiographically measurable disease not required
* Gemcitabine hydrochloride-refractory disease

  * Has undergone 1-3 prior therapies for locally advanced or metastatic disease with ≥ 1 regimen containing gemcitabine hydrochloride (alone or in combination with other agents)

    * Treatment given in the adjuvant setting (radiotherapy and/or chemotherapy, given either concurrently or systemically) does not count as prior therapy as long as progressive disease occurs > 6 months after completion of treatment
* No central nervous system (CNS) or brain metastases

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* International Normalized Ratio (INR) ≤ 1.5 (except in patients receiving full-dose warfarin)
* Bilirubin ≤ 2.0 mg/dL
* Creatinine ≤ 2.0 mg/dL
* AST or ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if documented liver metastases)
* Hemoglobin ≥ 9 g/dL (transfusion or epoetin alfa allowed)
* No contact lense use during and for 14 days after completion of study treatment
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* No history of other disease, metabolic dysfunction, or physical examination or clinical laboratory finding that contraindicates use of an investigational drug or precludes study compliance
* No history of serious systemic disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * Stroke within the past 6 months
  * Uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg on medication)
  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * Unstable symptomatic arrhythmia requiring medication

    * Chronic atrial arrhythmia (i.e., atrial fibrillation or paroxysmal supraventricular tachycardia) allowed
  * Peripheral vascular disease ≥ grade 2
* No significant traumatic injury within the past 28 days
* No proteinuria (defined as urine protein:creatinine ratio ≥ 1.0 at screening)
* No clinically significant impairment of renal function
* No serious, nonhealing wound, ulcer, or bone fracture
* No evidence of bleeding diathesis or coagulopathy
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months

PRIOR CONCURRENT THERAPY:

* More than 28 days since prior major surgery or open biopsy
* More than 7 days since prior fine-needle aspiration or core biopsy
* No prior antiangiogenesis agent (e.g., bevacizumab or an oral vascular endothelial growth factor receptor small molecule inhibitor) given together with an agent that disrupts epidermal growth factor receptor signaling (e.g., cetuximab or erlotinib hydrochloride) for locally advanced or metastatic pancreatic cancer

  * Prior treatment with either one of the above alone allowed
* More than 4 weeks since prior and no concurrent participation in another clinical trial
* No other concurrent antineoplastic or antitumor agents, including chemotherapy, radiotherapy, immunotherapy, or hormonal anticancer therapy
* No concurrent major surgery
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-02; Primary Completion 2009-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ko, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Result] Ko AH, Venook AP, Bergsland EK, Kelley RK, Korn WM, Dito E, Schillinger B, Scott J, Hwang J, Tempero MA. A phase II study of bevacizumab plus erlotinib for gemcitabine-refractory metastatic pancreatic cancer. Cancer Chemother Pharmacol. 2010 Nov;66(6):1051-7. doi: 10.1007/s00280-010-1257-5. Epub 2010 Feb 4. PMID 20130876
- [Result] Ko AH, Dito E, Schillinger B, et al.: A phase II study of bevacizumab (BEV) and erlotinib (ERL) in patients with gemcitabine (GEM)-refractory metastatic adenocarcinoma of the pancreas (PanCa). [Abstract] American Society of Clinical Oncology 2007 Gastrointestinal Cancers Symposium, 19 -21 January 2007, Orlando, Florida A-187, 2007.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at a single U.S. clinical site between March 2006 and December 2008
Groups:
- Bevacizumab Plus Erlotinib: Patients received bevacizumab 15 mg/kg as a 60-90 minute infusion every 21 days (representing one treatment cycle) and erlotinib 150 mg by mouth daily
Period: Overall Study
Arm/Group | Bevacizumab Plus Erlotinib
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab Plus Erlotinib
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 36
Number of prior lines of systemic therapy [Number; unit: Participants] — Patients must have received at least one, but no more than three, prior systemic therapies for advanced disease, at least one of which was gemcitabine based
  Participants
    1 Prior Line of Therapy | 24
    2 Prior Lines of Therapy | 9
    3 Prior Lines of Therapy | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate at 6 Months
Description: Number of participants alive at 6 months
Time Frame: 6 months
Population: All participants were followed for survival
Measure: Number; unit: participants
Arm/Group | Bevacizumab Plus Erlotinib
Number analyzed (Participants) | 36
participants | 8

2. Primary Outcome: Safety and Toxicity
Description: Treatment associated toxicities. Adverse event assessments were performed on day 1 of each treatment cycle and at the end of treatment; the longest duration of treatment was 7 cycles (x 3 weeks)
Time Frame: 21 weeks
Measure: Number; unit: participants
Arm/Group | Bevacizumab Plus Erlotinib
Number analyzed (Participants) | 36
participants
  Rash (Grades 1-3) | 26
  Diarrhea (Grades 1-3) | 9
  Hypertension (grade 3) | 4
  Gastrointestinal Bleeding (Grades 1 & 3) | 2
  Venous thromboembolic events (Grades 2-3) | 3
  Pulmonary embolism | 2
  Pancratogastic fistula | 1
  Suspected hemorrhage into intrapulmonic metastases | 1

3. Secondary Outcome: Objective Response as Measured by RECIST Criteria
Description: Participants experiencing objecting response, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 21 weeks
Measure: Number; unit: participants
Arm/Group | Bevacizumab Plus Erlotinib
Number analyzed (Participants) | 36
participants | 1

4. Secondary Outcome: Time to Tumor Progression
Description: Time to tumor progression (TTP) was defined as the time from initial therapy to the first objective documentation of tumor progression (for patients with measurable disease) or to the data of death, if death was ascribed to progression of disease.
Time Frame: from initial therapy to the first objective documentation of tumor progression
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Bevacizumab Plus Erlotinib
Number analyzed (Participants) | 36
Days | 40 [35 to 41]

5. Secondary Outcome: Proportion of Patients With ≥ 25% Decline in Serum CA19-9 Biomarker
Time Frame: 21 weeks
Population: Only patients with an elevated baseline CA19-9 (>2x ULN) were included in this analysis (n = 26).
Measure: Count of Participants; unit: Participants
Groups:
- Bevacizumab Plus Erlotinib Hydrochloride: A treatment cycle is 21 days:
  bevacizumab 15 mg/kg as a 60-90 min infusion once every 21 days, with erlotinib hydrochloride 150 mg by mouth daily
  bevacizumab
  erlotinib hydrochloride
  laboratory biomarker analysis
Arm/Group | Bevacizumab Plus Erlotinib Hydrochloride
Number analyzed (Participants) | 26
Participants | 4

ADVERSE EVENTS:
Time Frame: 21 weeks
Description: Participants were followed for adverse events while on study treatment; the longest duration on study was 7 cycles (x 3 weeks). Due to the severe illness of pancreatic cancer patients, the study did not collect AEs and SAEs unrelated to study treatment (due to disease).
Arm/Group | Bevacizumab Plus Erlotinib
Serious Adverse Events (participants affected / at risk) | 10/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Plus Erlotinib (N=36)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hypertension (Cardiac disorders) | 4 (4)
Venous Thromboembolic events (Vascular disorders) | 3 (3)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Plus Erlotinib (N=36)
Upper GI Bleed (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — "unexplained severe abdominal pain not related to disease progression"
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 25 (25)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Venous thromboembolic events (Vascular disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pancreatogastric fistula (Gastrointestinal disorders) | 1 (1)
Suspected hemorrhage into intrapulmonic metastases (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes